CLINICAL TRIAL: NCT04154319
Title: HPV Vaccination Among Daughters of Latina Immigrants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-120503007
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Cervical Cancer; Healthy Diet
Keywords: HPV vaccination; Healthy Eating; Latina immigrants
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Group randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Vaccination (Active Comparator): Mothers participated in educational/behavior change sessions to promote HPV vaccination among their 9-12 year old daughters
  Interventions: Behavioral: HPV Vaccination; Behavioral: Healthy Eating
- Healthy Eating (Active Comparator): Mothers and daughters participated in educational/behavior change sessions to promote healthy eating and appropriate nutrition label interpretation
  Interventions: Behavioral: Healthy Eating

INTERVENTIONS:
Behavioral: HPV Vaccination — Mothers assigned to this arm participated in educational/behavior change sessions to promote HPV vaccination among their unvaccinated 9-12 year old daughters
  Arms: HPV Vaccination
Behavioral: Healthy Eating — Mothers and daughters assigned to this arm received education on healthy eating and how to appropriately interpret nutrition labels

SUMMARY:
The overall goal of this study to promote HPV vaccine uptake among daughters of Latina immigrants between the ages of 9 and 12.

DETAILED DESCRIPTION:
Objective: Implementation and examination of the efficacy of a culturally relevant, community-based HPV vaccination intervention among daughters of Latina immigrants 9-12 years of age in Alabama.

Methods: Group-randomized controlled trial evaluating two interventions: 1) promotion of HPV vaccination and 2) promotion of healthy eating using "place of residence" as the unit of randomization. Between May 2013 and October 2017, forty locations with 317 mother-daughter dyads were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Latina immigrant
* Resident of selected randomization unit (place of residence)
* 18 years of age and older
* At least one HPV unvaccinated daughter between the ages of 9 and 12

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 634 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

PRIMARY OUTCOMES:
HPV vaccination among 9-12yo daughters of Latina immigrants | 7 months
  Daughters of mothers assigned to the HPV vaccination arm will more likely to complete the recommended HPV doses at 7-month follow-up than daughters of mothers assigned to the healthy eating arm.
Healthy eating among Latina immigrants and their 9-12 yo daughters | 7 months
  Mothers and daughters assigned to the healthy eating arm will be more likely to eat fried food less than once per week, consume at least three portions of fruit/vegetables per day and have less than one sweetened beverage per day at 7-months than mothers and daughters assigned to the HPV vaccination arm
Appropriate nutrition label interpretation among Latina immigrants mothers and 9-'12yo daughters | 7 months
  Mothers and daughters assigned to the healthy eating arm will be more likely to read nutrition labels sometimes/always and correctly interpret nutrition labels than mothers and daughters assigned to the HPV vaccination arm

REFERENCES:
- [Derived] Scarinci IC, Hansen B, Kim YI. A Cluster-Randomized Controlled Trial to Evaluate a Community-Based Healthy Eating and Nutrition Label Interpretation Intervention Among Latinx Immigrant Mothers and Their Daughters. J Community Health. 2021 Apr;46(2):313-323. doi: 10.1007/s10900-020-00885-x. PMID 32671515